CLINICAL TRIAL: NCT02120365
Title: Rapid Determination Of The Clinical Utility Of Perampanel For The Treatment Of Alcohol Dependence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Connecticut (Other); Yale University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Albert Arias, Associate Professor of Psychiatry, Virginia Commonwealth University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20014446; 1407014397 (Other: Yale University); R21AA026681 (NIH)
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Alcoholism
Keywords: Alcoholism; Heavy Drinking; Perampanel
MeSH Terms: conditions — Alcoholism | interventions — perampanel; Anticonvulsants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Perampanel 6mg (Experimental): Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg days prior to each test day, and then observed dosing moderate 6mg dose perampanel in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses [target Breath Alcohol Concentration (BrAc) =20mg%, 60mg%, and 100mg%] in a step-wise fashion.
  Interventions: Drug: Perampanel
- Placebo (Placebo Comparator): Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with placebo 7 days prior to each test day, and then observed dosing of placebo in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses [target Breath Alcohol Concentration (BrAc) =20mg%, 60mg%, and 100mg%] in a step-wise fashion.
  Interventions: Drug: Placebo
- Perampanel 10 mg (Experimental): Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg 7 days prior to each test day, and then observed dosing of high dose perampanel (10mg) in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses [target Breath Alcohol Concentration (BrAc) =20mg%, 60mg%, and 100mg%] in a step-wise fashion.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel is a noncompetitive (allosteric) antagonist of the AMPA-R that is well-absorbed (100% bioavailability), has good blood-brain-barrier penetration, and rapidly reaches peak plasma concentrations (1 hour). To date, there have been no clinical trials of AMPA-R antagonists (e.g., perampanel) for the treatment of alcoholism.
  Other Names: AMPA-R antagonist; anticonvulsant
  Arms: Perampanel 10 mg; Perampanel 6mg
Drug: Placebo — Placebo given in place of perampanel during the pre-treatment period and lab session days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether perampanel alters the response to alcohol for heavy drinkers. It is hypothesized that perampanel will reduce the rewarding and reinforcing properties of alcohol in the laboratory setting.

DETAILED DESCRIPTION:
The main goal of the proposed study is to determine whether the alpha-amino-3-hydroxy-5-methyl-4-isoxazoleproprionic acid receptor (AMPA-R) antagonist perampanel alters the response to ethanol (i.e., the rewarding and reinforcing effects) using a validated laboratory paradigm of intravenous (IV) ethanol infusion. Fifty non-treatment seeking heavy drinkers (NTSHDs), N=50, and twenty-five social drinkers (N=25) will undergo three test days each: once after receiving a placebo medication, once after receiving moderate dose perampanel, and once after receiving a higher dose of perampanel. This experiment is the first step in a series of expedient studies that will rapidly determine perampanel's potential as a treatment for alcohol dependence. If findings show perampanel reduces the rewarding and reinforcing properties of alcohol in the laboratory setting (in humans), it would provide a strong rationale for clinical treatment trials with this medication. This approach is innovative because it tests a highly novel AMPA-R antagonist for the treatment of alcoholism, and uses a state-of-the-art computer assisted IV alcohol pump infusion system (called CAIS) to reduce variability in blood alcohol concentrations, thus improving the data quality.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* between the ages of 21 and 55 years;
* Nontreatment-seeking Heavy Drinkers (NTSHDs)as defined above, and must have had at least 5 Standard Drinks (SD) in one day on at least some occasions in the past and been able to tolerate it without an adverse reaction
* generally medically and neurologically healthy on the basis of history, physical examination, Electrocardiogram, screening laboratory results (Complete Blood Count w/ differential, Thyroid Stimulating Hormone, Free-T4, Aspartate Transferase, Alanine Transferase, Gamma-Glutamyl Transferase, Blood Urea Nitrogen, creatinine, electrolytes, urinalysis, beta-Human Chorionic Gonadotropin). Individuals with Liver Function Tests (LFT) that are no more than 3 times above the normal levels will be included;
* women with a negative pregnancy test and not nursing, must be regularly using birth control
* negative breath alcohol at screening and on each test day;
* not taking any psychoactive medication or opioids (in past 30-days);
* are non-treatment seeking.

Exclusion Criteria:

* they need detoxification determined by a Clinical Institute Withdrawal Assessment (CIWA) score of >8 or have had a history of alcohol detoxification in the past;
* have been in treatment for an alcohol problem within the last 6 months, or if the severity of their alcohol problem based on the research physician's assessment warrants definitive treatment;
* meet criteria for Diagnostic Statistical Manual (DSM) -IV psychiatric and substance use disorder diagnosis (other than alcohol abuse/dependence, cannabis abuse/dependence and nicotine dependence; those diagnoses will be allowed; participants can be either smokers up to 1 pack per day or non-smokers) based on history and psychiatric evaluation that includes a structured diagnostic interview (Structured Clinical Interview for DSM-IV Axis I Disorders: SCID)
* unwillingness to remain alcohol-free 12 hours prior to test days;
* have a significant ongoing serious medical condition such as Diabetes Mellitus, liver disease (see above LFT guideline), renal disease (as evidenced by serum creatinine above our laboratory's reference limit of 1.7 mg/dL, or have a history of adverse reaction to IV placement/blood draw

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Arias, MD, Principal Investigator — Virginia CommonwealthUniversity
Locations (4):
- United States (4):
  - University of Connecticut, Farmington, Connecticut
  - Yale New Haven Hospital Research Unit, New Haven, Connecticut
  - West Haven Veterans Affairs, West Haven, Connecticut
  - Albert Arias, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: random assignment. Crossover
Groups:
- Placebo, Then Perampanel 6mg, Then Perampanel 10mg: Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg days prior to each test day, and then observed dosing moderate 6mg dose perampanel in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses [target Breath Alcohol Concentration (BrAC) =20mg%, 60mg%, and 100mg%] in a step-wise fashion.
  Perampanel: Perampanel is a noncompetitive (allosteric) antagonist of the alpha-amino-3-hydroxy-5-methyl-4-isoxazoleproprionic acid (AMPA)-Receptor that is well-absorbed (100% bioavailability), has good blood-brain-barrier penetration, and rapidly reaches peak plasma concentrations (1 hour). To date, there have been no clinical trials of AMPA-R antagonists (e.g., perampanel) for the treatment of alcoholism.
- Placebo, Then Perampanel 10mg, Then Perampanel 6mg; Perampanel 6mg, Then Placebo, Then Perampanel 10mg; Perampanel 6mg, Then Perampanel 10mg, Then Placebo; Perampanel 10mg, Then Perampanel 6mg, Then Placebo: Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg days prior to each test day, and then observed dosing moderate 6mg dose perampanel in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses [target BrAc (Breath Alcohol Concentration) =20mg%, 60mg%, and 100mg%] in a step-wise fashion.
  Perampanel: Perampanel is a noncompetitive (allosteric) antagonist of the AMPA-R that is well-absorbed (100% bioavailability), has good blood-brain-barrier penetration, and rapidly reaches peak plasma concentrations (1 hour). To date, there have been no clinical trials of AMPA-R antagonists (e.g., perampanel) for the treatment of alcoholism.
- Perampanel 10mg, Then Placebo, Then Perampanel 6mg: Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg 7 days prior to each test day, and then observed dosing of high dose perampanel (10mg) in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses (target BrAc=20mg%, 60mg%, and 100mg%) in a step-wise fashion.
  Perampanel: Perampanel is a noncompetitive (allosteric) antagonist of the AMPA-R that is well-absorbed (100% bioavailability), has good blood-brain-barrier penetration, and rapidly reaches peak plasma concentrations (1 hour). To date, there have been no clinical trials of AMPA-R antagonists (e.g., perampanel) for the treatment of alcoholism.
Period: Overall Study
Arm/Group | Placebo, Then Perampanel 6mg, Then Perampanel 10mg | Placebo, Then Perampanel 10mg, Then Perampanel 6mg | Perampanel 6mg, Then Placebo, Then Perampanel 10mg | Perampanel 6mg, Then Perampanel 10mg, Then Placebo | Perampanel 10mg, Then Perampanel 6mg, Then Placebo | Perampanel 10mg, Then Placebo, Then Perampanel 6mg
Started | 4 | 4 | 5 | 4 | 3 | 2
Completed | 4 | 4 | 3 | 0 | 3 | 0
Not Completed | 0 | 0 | 2 | 4 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 4 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Non-treatment seeking heavy drinkers- This is a crossover design. Subjects each completed at least one of the three dosages for a lab day.
Groups:
- Combined Group Crossover Study - Placebo/6mg/10mg: Crossover design with all participants completing three conditions. Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg days prior to each test day, and then observed dosing moderate 6mg dose perampanel in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses (target BrAc=20mg%, 60mg%, and 100mg%) in a step-wise fashion.
  Perampanel: Perampanel is a noncompetitive (allosteric) antagonist of the AMPA-R that is well-absorbed (100% bioavailability), has good blood-brain-barrier penetration, and rapidly reaches peak plasma concentrations (1 hour). To date, there have been no clinical trials of AMPA-R antagonists (e.g., perampanel) for the treatment of alcoholism.
Arm/Group | Combined Group Crossover Study - Placebo/6mg/10mg
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Biphasic Alcohol Effects Scale (BAES): Stimulant Subscale
Description: A 14-item scale with 7 items designed to assess stimulant effects from alcohol intoxication and 7 items developed to measure the sedative effects of alcohol. This scale was selected as a primary outcome measure because it is sensitive to the effect of alcohol. This outcome item reports the Stimulant Subscale results analyzed with mixed models. Each item can be scored a minimum of zero (0) or up to 10 with the 10 representing feeling more or the most intoxicated in that item's description (e.g., "excited"). The minimum score is 0 and the maximum score is 70. For the time frame, the values at different time points were combined (averaged) into a single value that represents the effect during the time interval of interest (12 to 110 minutes).
Time Frame: 98 minutes
Population: Non-treatment Seeking Heavy Drinkers of whom all participated in three separate lab days, each following a different dose of perampanel or placebo.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo Medication Dose: This is the mean effect of the placebo dose on BAES Stimulant Subscale
- Perampanel 6mg Dose: This is the mean score of the 6mg dose of perampanel on the BAES Stimulant Subscale
- Perampanel 10mg Dose: This is the effect of the mean of the perampanel 10mg dose on the BAES Stimulant Subscale
Arm/Group | Placebo Medication Dose | Perampanel 6mg Dose | Perampanel 10mg Dose
Number analyzed (Participants) | 14 | 17 | 15
score on a scale | 13.756 (2.747) | 14.053 (2.658) | 13.026 (2.816)
Statistical Analysis 1: Comparison: Placebo Medication Dose vs Perampanel 6mg Dose vs Perampanel 10mg Dose; Medication dose was a within-subjects factor (crossover design); Test type: Superiority; p = 0.867, Mixed Models Analysis; Mean Difference (Final Values) = 0.729, Standard Error of Mean 1.986 — Representing the high dose 10mg compared to the placebo 0mg dose

2. Primary Outcome: Biphasic Alcohol Effects Scale (BAES)- Sedative Subscale
Description: A 14-item scale with 7 items designed to assess stimulant effects from alcohol intoxication and 7 items developed to measure the sedative effects of alcohol. This scale was selected as a primary outcome measure because it is sensitive to the effect of alcohol. This entry item show the results for the sedative subscale evaluated in mixed models. Each item can be scored a minimum of zero (0) or up to 10 with the 10 representing feeling more or the most intoxicated in that item's description (e.g., "sedated"). The minimum score is 0 and the maximum score is 70. For the time frame, the values at different time points were combined (averaged) into a single value that represents the effect during the time interval of interest (12 to 110 minutes).
Time Frame: 98 minutes
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg days prior to each test day, and then observed dosing moderate 6mg dose perampanel in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses (target BrAc=20mg%, 60mg%, and 100mg%) in a step-wise fashion.
  Perampanel: Perampanel is a noncompetitive (allosteric) antagonist of the AMPA-R that is well-absorbed (100% bioavailability), has good blood-brain-barrier penetration, and rapidly reaches peak plasma concentrations (1 hour). To date, there have been no clinical trials of AMPA-R antagonists (e.g., perampanel) for the treatment of alcoholism.
- Perampanel 6mg: Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with placebo 7 days prior to each test day, and then observed dosing of placebo in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses (target BrAc=20mg%, 60mg%, and 100mg%) in a step-wise fashion.
  Placebo: Placebo given in place of perampanel during the pre-treatment period and lab session days.
- Perampanel 10 mg: Participants will have 3 test days each, 2 weeks apart, in a randomized order, following either pretreatment with daily perampanel 2mg 7 days prior to each test day, and then observed dosing of high dose perampanel (10mg) in the lab 1 hour before a one-time alcohol infusion . Each lab session occurs exactly a week after starting the medication for that round. The wash out period between lab test session phases will be 7-10 days. Subjects will receive 2 days of 2mg perampanel after each lab to taper down (included in the washout period). The next appointment will be brief at the start of the next phase, at which point the next week of low dose perampanel or placebo will be started. With the washout period and the 7 day taper of the next phase, the actual lab sessions will occur 14-17 days apart. All test days will involve administration of alcohol with the same 3 target doses (target BrAc=20mg%, 60mg%, and 100mg%) in a step-wise fashion.
  Perampanel: Perampanel is a noncompetitive (allosteric) antagonist of the AMPA-R that is well-absorbed (100% bioavailability), has good blood-brain-barrier penetration, and rapidly reaches peak plasma concentrations (1 hour). To date, there have been no clinical trials of AMPA-R antagonists (e.g., perampanel) for the treatment of alcoholism.
Arm/Group | Placebo | Perampanel 6mg | Perampanel 10 mg
Number analyzed (Participants) | 14 | 17 | 15
score on a scale | 4.624 (1.784) | 7.159 (1.649) | 10.263 (1.797)
Statistical Analysis 1: Comparison: Placebo vs Perampanel 6mg vs Perampanel 10 mg; mixed models, medication was a within-subjects factor; Test type: Superiority; p = 0.071, Mixed Models Analysis; Mean Difference (Final Values) = 5.514, Standard Error of Mean 3.038 — Representing the high dose 10mg compared to the placebo 0mg dose

3. Primary Outcome: Drug Effects Questionaire (DEQ)
Description: consists of four items that measure current alcohol effects: 'feel alcohol', 'feel high', 'like alcohol', and 'want more alcohol'. For the time frame, the values at different time points were combined (averaged) into a single value that represents the effect during the time interval of interest (12 to 110 minutes). There are five items on the scale with scores of 0 to 100, and the total score is used by averaging all five items, thus, the minimum total score on the scale is 0 and the maximum is 100. The lowest score 0 represents "not at all" or not experiencing any drug effects from alcohol, and 100 represents "extremely" experiencing alcohol effects.
Time Frame: 98 min
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo Medication Dose: This is the mean effect of the placebo dose on DEQ scale score
- Perampanel 6mg Dose: This is the mean score of the 6mg dose of perampanel on the DEQ scale score
- Perampanel 10mg Dose: This is the effect of the mean of the perampanel 10mg dose on the DEQ score
Arm/Group | Placebo Medication Dose | Perampanel 6mg Dose | Perampanel 10mg Dose
Number analyzed (Participants) | 14 | 17 | 15
score on a scale | 42.538 (3.379) | 40.619 (3.269) | 43.267 (3.442)
Statistical Analysis 1: Comparison: Placebo Medication Dose vs Perampanel 6mg Dose vs Perampanel 10mg Dose; mixed models; Test type: Superiority; p = 0.667, Mixed Models Analysis; Mean Difference (Final Values) = 0.729, Standard Error of Mean 2.905 — Representing the high dose 10mg compared to the placebo 0mg dose

4. Secondary Outcome: Alcohol Urge Questionnaire (AUQ)
Description: A valid eight-item Likert-type scale designed to assess acute alcohol craving. Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by averaging the item scores. Higher scores reflect greater craving. The minimum score is 7, and the maximum is 49. For the time frame, the values at different time points were combined (averaged) into a single value that represents the effect during the time interval of interest (12 to 110 minutes).
Time Frame: 98 min
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo Medication Dose: This is the mean effect of the placebo dose on Alcohol Urge Questionnaire
- Perampanel 6mg Dose: This is the mean score of the 6mg dose of perampanel on on Alcohol Urge Questionnaire
- Perampanel 10mg Dose: This is the effect of the mean of the perampanel 10mg dose on the on Alcohol Urge Questionnaire
Arm/Group | Placebo Medication Dose | Perampanel 6mg Dose | Perampanel 10mg Dose
Number analyzed (Participants) | 14 | 17 | 15
score on a scale | 16.481 (1.266) | 17.314 (1.177) | 18.723 (1.289)
Statistical Analysis 1: Comparison: Placebo Medication Dose vs Perampanel 6mg Dose vs Perampanel 10mg Dose; Test type: Superiority; p = 0.285, Mixed Models Analysis; Mean Difference (Final Values) = 2.242, Standard Error of Mean 1.393 — Representing the high dose 10mg compared to the placebo 0mg dose

5. Secondary Outcome: Side Effect Questionnaire (SEQ)
Description: This consists of a list of side effects associated with perampanel (e.g., fatigue, dizziness), rated from 0="none" to 4="severe". The mean for each subject across all items is included in each group/arm mean. The lowest score on the scale would be 0 and the maximum 4, as the mean across items is taken and not a sum. For the time frame, the values at different time points were combined (averaged) into a single value that represents the effect during the time interval of interest (12 to 110 minutes).
Time Frame: 98 minutes
Population: Non-Treatment Seeking Heavy Drinkers
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo Medication Dose; Perampanel 6mg Dose; Perampanel 10mg Dose: This is the mean effect of the placebo dose on the Side Effect Questionnaire
Arm/Group | Placebo Medication Dose | Perampanel 6mg Dose | Perampanel 10mg Dose
Number analyzed (Participants) | 14 | 17 | 15
score on a scale | 0.895 (.294) | .992 (.261) | 1.13 (.280)
Statistical Analysis 1: Comparison: Placebo Medication Dose vs Perampanel 6mg Dose vs Perampanel 10mg Dose; Mixed Models; Test type: Superiority; p = .843, Mixed Models Analysis; Mean Difference (Final Values) = .235, Standard Error of Mean .408 — Representing the high dose 10mg compared to the placebo 0mg dose

6. Secondary Outcome: Profile of Mood States (POMS) 2 Short Version Total Score
Description: The Profile of Mood States (POMS) 2 short version contains a subset of 35 items from the full-length versions. This subset comprises those five items on full version POMS scale that exhibited good item-total correlations and best predicted their respective scale scores, this is a TOTAL score Representing total mood disturbance. For the time frame, the values at different time points were combined (averaged) into a single value that represents the effect during the time interval of interest (12 to 110 minutes). The minimum is 0 and the maximum is 100 with higher numbers indicating greater mood disturbance.
Time Frame: 98 minutes
Population: Nontreatment-seeking Heavy Drinkers (NTSHDs)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo Medication Dose; Perampanel 6mg Dose; Perampanel 10mg Dose: This is the mean effect of the placebo dose on the Profile of Mood States (POMS) 2
Arm/Group | Placebo Medication Dose | Perampanel 6mg Dose | Perampanel 10mg Dose
Number analyzed (Participants) | 14 | 17 | 15
score on a scale | 20.25 (1.490) | 21.75 (1.335) | 20.619 (1.533)
Statistical Analysis 1: Comparison: Placebo Medication Dose vs Perampanel 6mg Dose vs Perampanel 10mg Dose; We report the main effect of dose on the outcome measure; Test type: Superiority; p = .691, Mixed Models Analysis; Mean Difference (Final Values) = .369, Standard Error of Mean 2.07 — Representing the high dose 10mg compared to the placebo 0mg dose

ADVERSE EVENTS:
Time Frame: 40 days of participation
Arm/Group | Placebo | Perampanel 6mg | Perampanel 10 mg
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 4/22 | 1/22 | 4/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Perampanel 6mg (N=22) | Perampanel 10 mg (N=22)
nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) — nausea/vomiting
IV site bruising/thrombosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) — Intravenous access site side effect
Viral cold symptoms (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02120365/Prot_SAP_002.pdf
  • Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT02120365/ICF_003.pdf